CLINICAL TRIAL: NCT04559867
Title: Fistulotomy as the Primary Cannulation Technique for All Patients Undergoing ERCP: A Randomized, Controlled Trial
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: slower than expected recruitment
Sponsor: Lawrence Charles Hookey (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Director, Endoscopy, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6029074
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Biliary Tract Diseases
Keywords: Needle Knife Fistulotomy; Sphincterotomy; Post-ERCP pancreatitis
MeSH Terms: conditions — Biliary Tract Diseases | interventions — Sphincterotomy

STUDY DESIGN:
Intervention Model Description: During the procedure, the study doctor will evaluate the participant's anatomy to determine if both approaches are possible to safely perform. If both approaches are assessed as safe to perform, then the participant will be randomly assigned (like the toss of a coin) to one approach. If the study doctor is unable to gain access using the approach the patient is initially assigned to, then they will switch approaches and use the other approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle Knife Fistulotomy (Active Comparator): The study doctor will gain access to the bile ducts using the cutting technique called a needle knife fistulotomy. When using this technique, the study doctor makes a cut directly into the bile duct.
  Interventions: Procedure: Needle knife fistulotomy
- Sphincterotomy (Active Comparator): The study doctor will gain access to the bile ducts using the cutting technique called a sphincterotomy. Using this method, a heated metal wire cuts the opening to the bile duct after a wire has been passed into it.
  Interventions: Procedure: Sphincterotomy

INTERVENTIONS:
Procedure: Needle knife fistulotomy — A needle knife fistulotomy uses a tiny knife to cut directly into the ampulla to gain access to the biliary system in patients undergoing ERCP.
  Arms: Needle Knife Fistulotomy
Procedure: Sphincterotomy — A sphincterotomy uses a heated metal wire to cut the opening to the bile duct after a wire has been passed into it.
  Arms: Sphincterotomy

SUMMARY:
Participants in this study will be undergoing a procedure called an endoscopic retrograde cholangiopancreatography (ERCP). This procedure is most commonly performed to help treat conditions affecting specific areas of the digestive system called the pancreas and bile ducts.

Patients will consent to allow the study physician to access these areas of the digestive system by either making a cut called a needle-knife fistulotomy or a sphincterotomy.

DETAILED DESCRIPTION:
The ERCP procedure enables the study doctor to examine regions of the digestive system called the pancreas and bile ducts. After a patient is sedated, a bendable tube with a light (called an endoscope), is inserted through the mouth and into the digestive system. Within the digestive system, the doctor is able to identify the opening to where the gallbladder drains into the small bowel called the ampulla. Using the endoscope, a small plastic tube is then placed in the opening and dye (also called contrast material) is injected into the bile duct (area where bile leaves the liver). X-ray pictures can then be taken to provide further information to the doctor.

During the procedure, it is necessary to make a cut to enlarge the opening to allow easier removal of stones from the bile duct or to place plastic tubes (stents) in the bile duct. To make this cut, there are two different approaches that the doctor can take:

1. The standard way of making the cut is referred to as a "sphincterotomy". Using this method, a heated metal wire cuts the opening to the bile duct after a wire has been passed into it.
2. The second way of making the cut is referred to as a "pre-cut". There are various types of "pre-cut" techniques; the technique being evaluated in this study is called the "needle knife fistulotomy". When using this technique, the doctor makes a cut directly into the bile duct using a tiny knife called a "needle knife".

Currently, the doctor determines which cutting technique to use. The decision is entirely up to the individual doctor.

The purpose of this study, called a randomized, controlled trial, is to compare the safety and effectiveness of the two different approaches to the ERCP.

This type of study involves a large number of participants and the results may answer the question as to which approach should be used for patients having the ERCP procedure. The results may change the standard way that doctors conduct this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, greater than, or equal to 18 years of age, with an intact sphincter undergoing ERCP by at Kingston Health Sciences Center for therapeutic purposes who can provide informed consent. This includes patients who have confirmed choledocholithiasis on imaging and those who have a high suspicion of it based on imaging and lab values. Patients with and without a high suspicion for cholangitis will be eligible for the study. Other indications include: other benign biliary duct diseases including strictures, primary sclerosing cholangitis and Mirizzi's syndrome requiring biliary decompression. Furthermore, patients with suspected diagnosis of biliary leak following cholecystectomy will also be considered for enrollment in this study.
2. Ability to read and understand the English language,
3. Ability to follow-up in a reliable manner.

Exclusion Criteria:

1. Bleeding disorder (Von Willebrand disorder, platelet count <100 000, or INR >1.5),
2. Therapeutic level anticoagulation with low molecular weight heparin (LMWH), warfarin, or a direct-acting oral anticoagulant (DOAC),
3. P2Y12 inhibitors not held for 5 days prior to the procedure,
4. Prior biliary sphincterotomy,
5. Concurrent pancreatitis (with inability to tolerate oral intake and requiring pain management),
6. Altered upper GI tract anatomy (e.g. prior gastric bypass surgery such as Roux-en-Y or Billroth 2 gastrojejunostomy),
7. Inability to achieve adequate sedation,
8. Evidence of malignant infiltration of the ampulla or peri-ampullary area,
9. Pregnancy,
10. Operator inability to access and identify intra-duodenal portion of the bile duct,
11. Presumptive diagnosis of sphincter of Oddi dysfunction,
12. Inability to access intraduodenal segment due to altered anatomy (eg. ampulla within deep diverticulum),
13. Requirement for pancreatogram or pancreatic intervention,
14. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | Up to 7 days
  The primary objective to be examined is the incidence of post-ERCP pancreatitis.

SECONDARY OUTCOMES:
Cannulation Success Rate | Day 0
  Rate of successful cannulation of the common bile duct, with technical success determined by a cholangiogram.
Inspection Time | Day 0
  Inspection time of the ampulla, defined as the visualization of the ampulla to the appearance of the needle knife or sphinctertome.
Time to successful cannulation | Day 0
  For the sphincterotomy group, time to successful cannulation is defined as time of endoscopic visualization of the sphinctertome on the screen to contact with the papilla orifice. For the NKF group, this is defined as the time of endoscopic visualization of the metal point of the needle knife on the screen to successful cannulation of the common bile duct as evident by the cholangiogram or wire advancement into the common bile duct.
Total procedure time | Day 0
  Total procedure time is measured for completed procedures from the time of esophageal intubation to the time of scope withdrawal from the patient mouth.
Ampullary morphology | Day 0
  The type of ampulla, as determined by the study doctor.
Difficulty of cannulation | Day 0
  Difficulty of cannulation, as graded on a 3-point scale, based on the study doctor's subjective opinion.
Incidence of complications | Up to 7 days
  Incidence of complications, notably intraprocedural bleeding that required intervention, delayed or sustained bleeding requiring transfusion or repeat endoscopy, and immediate or delayed perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bechara, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davee T, Garcia JA, Baron TH. Precut sphincterotomy for selective biliary duct cannulation during endoscopic retrograde cholangiopancreatography. Ann Gastroenterol. 2012;25(4):291-302. PMID 24714256
- [Background] Robison LS, Varadarajulu S, Wilcox CM. Safety and success of precut biliary sphincterotomy: Is it linked to experience or expertise? World J Gastroenterol. 2007 Apr 21;13(15):2183-6. doi: 10.3748/wjg.v13.i15.2183. PMID 17465498
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Background] Andrade-Davila VF, Chavez-Tostado M, Davalos-Cobian C, Garcia-Correa J, Montano-Loza A, Fuentes-Orozco C, Macias-Amezcua MD, Garcia-Renteria J, Rendon-Felix J, Cortes-Lares JA, Ambriz-Gonzalez G, Cortes-Flores AO, Alvarez-Villasenor Adel S, Gonzalez-Ojeda A. Rectal indomethacin versus placebo to reduce the incidence of pancreatitis after endoscopic retrograde cholangiopancreatography: results of a controlled clinical trial. BMC Gastroenterol. 2015 Jul 21;15:85. doi: 10.1186/s12876-015-0314-2. PMID 26195123
- [Background] Buxbaum J, Yan A, Yeh K, Lane C, Nguyen N, Laine L. Aggressive hydration with lactated Ringer's solution reduces pancreatitis after endoscopic retrograde cholangiopancreatography. Clin Gastroenterol Hepatol. 2014 Feb;12(2):303-7.e1. doi: 10.1016/j.cgh.2013.07.026. Epub 2013 Aug 3. PMID 23920031
- [Background] Shaygan-Nejad A, Masjedizadeh AR, Ghavidel A, Ghojazadeh M, Khoshbaten M. Aggressive hydration with Lactated Ringer's solution as the prophylactic intervention for postendoscopic retrograde cholangiopancreatography pancreatitis: A randomized controlled double-blind clinical trial. J Res Med Sci. 2015 Sep;20(9):838-43. doi: 10.4103/1735-1995.170597. PMID 26759569
- [Background] Cavallini G, Tittobello A, Frulloni L, Masci E, Mariana A, Di Francesco V. Gabexate for the prevention of pancreatic damage related to endoscopic retrograde cholangiopancreatography. Gabexate in digestive endoscopy--Italian Group. N Engl J Med. 1996 Sep 26;335(13):919-23. doi: 10.1056/NEJM199609263351302. PMID 8786777
- [Background] Manes G, Ardizzone S, Lombardi G, Uomo G, Pieramico O, Porro GB. Efficacy of postprocedure administration of gabexate mesylate in the prevention of post-ERCP pancreatitis: a randomized, controlled, multicenter study. Gastrointest Endosc. 2007 Jun;65(7):982-7. doi: 10.1016/j.gie.2007.02.055. PMID 17531632
- [Background] Andriulli A, Clemente R, Solmi L, Terruzzi V, Suriani R, Sigillito A, Leandro G, Leo P, De Maio G, Perri F. Gabexate or somatostatin administration before ERCP in patients at high risk for post-ERCP pancreatitis: a multicenter, placebo-controlled, randomized clinical trial. Gastrointest Endosc. 2002 Oct;56(4):488-95. doi: 10.1067/mge.2002.128130. PMID 12297762
- [Background] Andriulli A, Solmi L, Loperfido S, Leo P, Festa V, Belmonte A, Spirito F, Silla M, Forte G, Terruzzi V, Marenco G, Ciliberto E, Sabatino A, Monica F, Magnolia MR, Perri F. Prophylaxis of ERCP-related pancreatitis: a randomized, controlled trial of somatostatin and gabexate mesylate. Clin Gastroenterol Hepatol. 2004 Aug;2(8):713-8. doi: 10.1016/s1542-3565(04)00295-2. PMID 15290665
- [Background] Yuhara H, Ogawa M, Kawaguchi Y, Igarashi M, Shimosegawa T, Mine T. Pharmacologic prophylaxis of post-endoscopic retrograde cholangiopancreatography pancreatitis: protease inhibitors and NSAIDs in a meta-analysis. J Gastroenterol. 2014 Mar;49(3):388-99. doi: 10.1007/s00535-013-0834-x. Epub 2013 May 30. PMID 23720090
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Katsinelos P, Gkagkalis S, Chatzimavroudis G, Beltsis A, Terzoudis S, Zavos C, Gatopoulou A, Lazaraki G, Vasiliadis T, Kountouras J. Comparison of three types of precut technique to achieve common bile duct cannulation: a retrospective analysis of 274 cases. Dig Dis Sci. 2012 Dec;57(12):3286-92. doi: 10.1007/s10620-012-2271-8. Epub 2012 Jun 20. PMID 22714730
- [Background] Sundaralingam P, Masson P, Bourke MJ. Early Precut Sphincterotomy Does Not Increase Risk During Endoscopic Retrograde Cholangiopancreatography in Patients With Difficult Biliary Access: A Meta-analysis of Randomized Controlled Trials. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1722-1729.e2. doi: 10.1016/j.cgh.2015.06.035. Epub 2015 Jul 2. PMID 26144018
- [Background] Ayoubi M, Sansoe G, Leone N, Castellino F. Comparison between needle-knife fistulotomy and standard cannulation in ERCP. World J Gastrointest Endosc. 2012 Sep 16;4(9):398-404. doi: 10.4253/wjge.v4.i9.398. PMID 23125897
- [Background] Jin YJ, Jeong S, Lee DH. Utility of needle-knife fistulotomy as an initial method of biliary cannulation to prevent post-ERCP pancreatitis in a highly selected at-risk group: a single-arm prospective feasibility study. Gastrointest Endosc. 2016 Nov;84(5):808-813. doi: 10.1016/j.gie.2016.04.011. Epub 2016 Apr 19. PMID 27102829
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Early precut fistulotomy for biliary access: time to change the paradigm of "the later, the better"? Gastrointest Endosc. 2014 Oct;80(4):634-641. doi: 10.1016/j.gie.2014.03.014. Epub 2014 May 6. PMID 24814775
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Derived] Hookey L, Rai M, Bechara R. Fistulotomy versus standard cannulation as the primary technique for all patients undergoing ERCP with a native papilla: a protocol for a single center randomized controlled trial. Trials. 2022 Feb 16;23(1):153. doi: 10.1186/s13063-022-06084-4. PMID 35172872